CLINICAL TRIAL: NCT00329706
Title: Early and Long-Term Value of Imaging Brain Metabolism
Brief Title: Metabolic Cerebral Imaging in Incipient Dementia (MCI-ID)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel H. Silverman, Professor, Medical and Molecular Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 02-10-079, 03-04-026
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Dementia
Keywords: mild cognitive impairment; Alzheimer's disease; dementia; FDG; PET
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental arm will have an immediate release of the PET report
  Interventions: Procedure: FDG-PET brain scan
- 2 (Active Comparator): Active Comparator arm will have a delayed release of 2 years
  Interventions: Procedure: FDG-PET brain scan

INTERVENTIONS:
Procedure: FDG-PET brain scan — The difference in the two arms' interventions is the time at which the FDG-PET brain scan information is available for the subjects' managing physicians. Experimental arms will have an immediate release of the PET report, while the Active Comparator arms will have a delayed release of 2 years.
  Other Names: [F-18]FDG PET brain scan administered once to both arms

SUMMARY:
A brain PET scan is recognized as "reasonable and necessary" for some patients with "a recently established diagnosis of dementia" (Centers for Medicare and Medicaid Services, Decision Memo CAG-00088R, 2004), but evidence is less clear for patients having less severe cognitive problems. A substantial portion of such patients will develop Alzheimer's disease and other forms of dementia, which affect millions of people in the U.S., costing us over $100 billion annually. This project employs a prospective randomized protocol to determine whether PET scanning can help distinguish those patients with early Alzheimer's changes in their brains from those having other causes of cognitive impairment more accurately than is done with current clinical practices alone, and lead to earlier, more effective therapies which extend patients' abilities to think and function independently.

DETAILED DESCRIPTION:
People experiencing mild cognitive changes represent an epidemiologically major segment of the geriatric patient population. In the present proposal, we aim to measure how knowledge of cerebral metabolic information 1) influences working diagnoses and management of patients being evaluated for symptoms of early cognitive decline, and 2) impacts upon long-term clinical outcomes, particularly of subjects having metabolic patterns consistent with presence of Alzheimer's disease (AD)-like changes in their brains. A total of 710 patients suffering from documentable decline of cognitive function in the absence of overt dementia will be studied at nine U.S. institutions with extensive experience and infrastructure in place for the evaluation of Alzheimer's disease and related disorders, and for neuroimaging. In this prospective, investigation, subjects will undergo baseline neuropsychologic testing and neuroimaging with MRI and FDGPET. PET scan reports will be sealed and randomized with respect to whether they are released to patients' managing physicians at the time of interpretation, or two years after the time that scanning is performed.

Working diagnoses of managing physicians will be recorded, as will the treatment decisions made by the managing physicians and their patients. Cognitive abilities, functional status, utilization of healthcare resources, and other clinical and social contact parameters will be assessed every six months. Our major hypotheses are that among patients whose PET results are immediately conveyed to their referring physicians, diagnoses and management plans will be positively affected, leading to more effective utilization of healthcare resources and to maintenance of cognitive and functional abilities at a higher level. This project will also provide a rich source of data that can be used to address questions outside of its major focus (e.g., prognostic accuracy of volumetric MRI data used instead of, or in conjunction with, FDG-PET data; incremental predictive value of applying statistically parameterizing and/or quantifying software tools to imaging data).

ELIGIBILITY:
Inclusion Criteria:

* Cognitive deficit and/or personality change is present, as observable by physician and/or close contact(s) of the patient; or in the absence of this, the patient provides a clear history of decline which the patient's physician deems to be reliable.
* If history or neurologic exam reveals findings suspicious for stroke, tumor, bleed, ictal activity, or hydrocephalus, then CT/MRI and appropriate neurological or neurosurgical consultation must have been obtained.
* Standard history, physical, and laboratory screen have been performed to identify possible presence of depression, substance abuse, malnourishment, medication effects and interactions, cardiopulmonary compromise, electrolyte/calcium imbalance, anemia, hypoxemia, infection, thyroid dysfunction, renal dysfunction, hepatic dysfunction, or glucose dysregulation.
* Any positive findings revealed in 2) or 3) above have been appropriately treated, wherever possible, but cognitive/behavioral deficit persists post-therapy.

Exclusion Criteria:

* Subjects under age 65 will not be recruited, in order to enhance the clinical relevance of the project by focusing on the age groups in whom serious concerns about early signs and symptoms of senile onset dementia are most typically emerging.
* Overt dementia, as discussed above.
* Cognitive dysfunction has impaired subject's ability to perform activities of daily living.
* Present or past history of thyroid disease (due to effects of both the disease and thyroid hormone replacement therapy on brain metabolism that we and others have begun to identify, but which remain incompletely characterized.)
* Claustrophobia or metal in body or other condition that would preclude PET or MRI from being acquired, or visual, auditory or motor deficits that would preclude accurate neuropsychological testing.
* Cholinesterase inhibition therapy already initiated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 710 (Actual)
Dates: Start 2006-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in neuropsychological (cognitive,functional) test results | baseline and 2 years
utilization of healthcare resources | baseline and 2 years
PET results, compared with working diagnoses made before and after time of PET | baseline and up to 2 years
rates of prescription of AD-specific therapies | baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Silverman, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (9):
- United States (9):
  - Mayo Clinic, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Santa Monica-UCLA Medical Center, Santa Monica, California
  - Gene E. Myers Cardiac and Vascular Consultants, Sarasota, Florida
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - University of Buffalo, Buffalo, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah